CLINICAL TRIAL: NCT01814917
Title: A Multi-centre, Flexible Dose, Parallel Group, Open-label, Active Control (Calcium-based Phosphate Binder), Long-term Extension Study Evaluating the Efficacy, Safety and Tolerability of Colestilan (MCI-196) in Paediatric Subjects With Hyperphosphataemia and With Either Chronic Kidney Disease Stage 5 on Dialysis or Chronic Kidney Disease Stages 3b to 5 Not on Dialysis
Brief Title: Long-term Extension Study of MCI-196
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study has been terminated because of insufficient patient recruitment.
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCI-196-E15
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Kidney Disease; Dialysis; Hyperphosphatemia; Paediatric
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia | interventions — cholebine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MCI-196 (Flexible dose) (Experimental): MCI-196 BSA eq 3g, 6g, 9g, 12g or 15g
  Interventions: Drug: colestilan
- CBPB (Active Comparator): Calcium-based P binder
  Interventions: Drug: CBPB

INTERVENTIONS:
Drug: colestilan — body surface area equivalent (BSAeq) 3 g/day, 6 g/day, 9 g/day, 12 g/day or 15 g/day
  Other Names: BindRen
  Arms: MCI-196 (Flexible dose)
Drug: CBPB
  Arms: CBPB

SUMMARY:
The Primary Objectives of this study are to assess the long-term efficacy of treatment with colestilan (MCI-196) (including combination therapy) and to assess the long-term safety of treatment with colestilan (MCI-196) (including combination therapy).

DETAILED DESCRIPTION:
This study has been terminated because of insufficient patient recruitment. There were no safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* The subject and/or parent(s)/guardian(s) must be capable of providing informed consent, and assent when applicable, in agreement with regional requirements.
* The subject has completed either of the short-term studies, MCI-196-E14 or MCI-196-E16

or

* The subject has been withdrawn from MCI-196-E14, but is eligible to enter this study according to the following rules, as defined in MCI-196-E14:

  * Hyperphosphataemia: Subjects who experienced hyperphosphataemia, defined as any increase in serum phosphorus [P] levels above the age-related upper limit of normal(ULN) on two consecutive occasions, and was withdrawn by the Investigator in order to proceed to this study, where flexible dosing with colestilan (MCI-196) is available. Subjects withdrawn from MCI-196-E14 due to hyperphosphataemia may only enter this study after Week 6 of the short-term study, following two consecutive out-of-range P values (one obtained at Week 3 and one obtained at Week 6). After Week 6, subjects meeting the above criteria may enter this study at any time (the two consecutive out-of-range P values having been obtained any time after Week 6 from a scheduled or unscheduled visit).
  * Hypercalcaemia: Subjects treated with CBPB and experiencing hypercalcaemia may be withdrawn from the short-term study at the discretion of the Investigator in order to proceed to this study at any time, where flexible dosing with colestilan (MCI-196) is available.

Exclusion Criteria:

* The subject has current clinically significant medical co-morbidities, which may substantially compromise subject safety, or expose them to undue risk, or interfere significantly with study procedures and which, in the opinion of the Investigator, make the subject unsuitable for inclusion in the study (e.g., the subject currently has or has had a history of seizure disorders, dysphagia, swallowing disorders, predisposition to or current bowel obstruction, ileus or severe gastrointestinal [GI] disorders such as chronic or severe constipation [as judged by the Investigator], intestinal stenosis, intestinal diverticulum, sigmoid colitis, GI ulcers, current or a history of GI bleeding, or major GI tract surgery).
* The subject is expected to receive immunosuppressant treatment during the course of the study.
* The subject is considered unstable on his/her current treatment for CKD within one month prior to enrolment (e.g., subjects starting treatment with vitamin D or its analogues, or other agents/procedures that may influence bone mineral metabolism [i.e., serum P and calcium (Ca) levels]).
* The subject is considered to be non-compliant with study procedures in the opinion of the Investigator.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Proportion of responders (responders are defined as subjects demonstrating serum P levels ≤1.5 SD above the KDOQI 2008 age-related mean value) | 52 weeks
  Kidney Disease Outcomes Quality Initiative (KDOQI)

SECONDARY OUTCOMES:
Mean absolute change in efficacy laboratory parameters (i.e.,P, Ca, Ca P ion product [CaxP], intact parathyroid hormone [iPTH], serum glucose, glycosylated haemoglobin [HbA1c], and uric acid) | 52 weeks
Mean percentage change in other efficacy laboratory parameters (i.e., lipid parameters [low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C), total cholesterol, and triglycerides (TG)]) | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational site, London, United Kingdom